CLINICAL TRIAL: NCT00313768
Title: A Randomized Phase 2 Trial Of Paclitaxel, Carboplatin And Bevacizumab With Or Without PF-3512676 As First-Line Treatment Of Patients With Advanced Nonsquamous Non-Small Cell Lung Cancer
Brief Title: Randomized Ph 2 Trial Of Paclitaxel/Carboplatin /Bevacizumab + PF-3512676 And P/C/B Alone In Advanced Nonsquamous NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Termination Reason in Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501003
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced carcinoma, non-small cell lung, Phase II, paclitaxel, Taxol, carboplatin, Paraplatin, bevacizumab, Avastin, PF-3512676, immunotherapy, immunomodulator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Bevacizumab; ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): Standard of care chemotherapy
  Interventions: Drug: paclitaxel + carboplatin + bevacizumab
- A (Experimental): Standard of care chemotherapy plus experimental intervention (PF-3512676)
  Interventions: Drug: carboplatin + paclitaxel + bevacizumab + PF-3512676

INTERVENTIONS:
Drug: paclitaxel + carboplatin + bevacizumab — paclitaxel 200 mg/m2 intravenously Day 1 of each 21 day cycle x 6 cycles
  Other Names: Taxol; Paraplatin
  Arms: B
Drug: carboplatin + paclitaxel + bevacizumab + PF-3512676 — carboplatin AUC 6 intravenously on Day 1 of each 21 day cycle x 6 cycles
  Other Names: Paraplatin; Taxol; Avastin
  Arms: A

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with paclitaxel, carboplatin and bevacizumab as first-line treatment in patients with locally advanced or metastatic nonsquamous non-small cell lung cancer

DETAILED DESCRIPTION:
PF-3512676 dosing was stopped 21 June 2007 when Pfizer decided to stop the administration of PF-3512676 in all trials which combined PF-3512676 with cytotoxic chemotherapy. the decision was made subsequent to DSMC recommendation to close two phase III randomized trials in non-small cell lung cancer which also combined PF-3512676 with cytotoxic chemotherapy, citing lack of efficacy concerns as the primary reason with safety issues (sepsis, thrombocytopenia) also contributing to the decision. Subjects were allowed to complete standard of care treatment/survival follow-up. Data collection was completed on 22 May 2008.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Stage IIIb with pleural effusion or Stage IV nonsquamous non-small cell lung cancer
* ECOG Performance Status 0-1
* Measurable disease per RECIST criteria

Exclusion Criteria:

* Squamous cell, small cell, or carcinoid lung cancer
* CNS metastasis
* Pre-existing autoimmune or antibody mediated disease
* Prior systemic treatment for NSCLC with chemo, immunotherapy, biologics, or investigation drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 110 Events

SECONDARY OUTCOMES:
Time to Tumor Progression | End of treatment
Overall Objective Response Rate | Time of progressive disease
Duration of Response | Time of progression
Overall Survival | Time of death
Overall safety profile | 28 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Bessemer, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Cocoa Beach, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Rockledge, Florida
  - Pfizer Investigational Site, Titusville, Florida
  - Pfizer Investigational Site, Valdosta, Georgia
  - Pfizer Investigational Site, Joliet, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Pollocksville, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, San Marcos, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501003&StudyName=Randomized%20Ph%202%20Trial%20Of%20Paclitaxel/Carboplatin%20/Bevacizumab%20+%20PF-3512676%20And%20P/C/B%20Alone%20In%20Advanced%20Nonsquamous%20NSCLC%0A